CLINICAL TRIAL: NCT07243756
Title: A Pilot Proof of Concept Study, Single-center, Open-label Study to Assess the Safety and Efficacy of an Ingestible Pill for Gut Microbiome Sampling in Healthy Humans
Brief Title: Gut Microbiome Pill
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-00116
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: microbiome; microbiota; microbiome sampling pill

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microbiome sampling (Experimental): Participants will ingest one single 3D-printed pill and monitor for the pill in their stool over the next 4 days using a metal detection device. Upon detection participants will collect a sample of the stool and the pill.
  Interventions: Device: 3D-printed ingestible pill

INTERVENTIONS:
Device: 3D-printed ingestible pill — The pill consists of a microporous architecture specifically designed to trap bacteria. The pill contains a ferrous (iron) ball for detection with a metal detection device and passes naturally and passively through the GI tract.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a 3D-printed ingestible pill designed to sample microbiota from the GI tract, focusing on the ability to collect data also from the small intestine. The study also aims to assess ease of use and transit time.

DETAILED DESCRIPTION:
This is a prospective, open-label pilot study designed to evaluate the safety and efficacy of a 3D-printed ingestible pill for microbiome sampling throughout the gastrointestinal (GI) tract, with a specific advantage in being able to sample bacteria from the small intestine. The study will enroll 10 participants, each ingesting the pill. Participants will use a metal detection device to identify the pill in their stool. Upon detection, participants will collect the stool sample and send it to the lab, where the pill will be extracted. Both the pill and stool samples will undergo 16S rRNA sequencing to profile the microbiome. The study will take approximately 4 days per participant

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18-65.
2. Willing and able to provide informed consent.
3. Able and willing to comply with study procedures, including pill ingestion, stool collection, follow and record dietary instructions, and fill questionnaires.

Exclusion Criteria:

1. History of gastrointestinal diseases (e.g., Crohn's disease, irritable bowel syndrome, small intestinal bacterial overgrowth).
2. History of abdominal surgery that may impact gastrointestinal function (e.g., bowel resection, bariatric surgery).
3. Known allergies or intolerances to medical devices or ingestible capsules.
4. Recent antibiotic use (within 3 months) that may affect gut microbiome results.
5. Use of medications that alter GI motility such as laxatives or prokinetics.
6. Known anatomical abnormalities or strictures in the GI tract that increase the risk of obstruction.
7. Pregnant, planning pregnancy or breastfeeding, since pregnancy and breastfeeding affect the microbiome, Exclusion of pregnancy will be confirmed by the date of the last menstrual period.
8. Participation in another investigational trial within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who successfully passed the pill through the GI tract without causing any adverse effects such as GI discomfort, obstruction, or other complications | Pill retrieval (up to 4 days)
  Participants will be asked to report any subsequent events to the study team. Adverse Events (AEs) will be collected through solicited questions (e.g., "Have you experienced any discomfort after ingesting the pill?") and unsolicited reports from participants. All events will be categorized, and severity will be graded.
Number of samples that accurately represents bacterial populations in the small intestine, as well as the entire GI tract, when compared to stool samples | Pill retrieval (up to 4 days)
  Outcome is evaluated using 16S ribosomal RNA (rRNA) sequencing to compare microbial diversity and the presence of specific bacterial taxa between the pill and stool samples.

SECONDARY OUTCOMES:
Time taken for the pill to pass through the GI tract | From ingestion until pill retrieval (up to 4 days)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Gross, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: seth.gross@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to seth.gross@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.